CLINICAL TRIAL: NCT01635829
Title: A Phase I, Open-label, Randomized, 2-panel, Sequential Treatment Study in Healthy Subjects to Investigate the Potential Pharmacokinetic Interactions Between Multiple Doses of Phenytoin or Carbamazepine and Telaprevir at Steady-state
Brief Title: A Study to Investigate the Potential Pharmacokinetic Interactions Between Phenytoin or Carbamazepine and Telaprevir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Infectious Diseases BVBA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100830; VX-950HPC1002 (Other: Janssen Infectious Diseases BVBA); 2012-001411-23 (EudraCT Number)
Record Dates: First submitted 2012-07-04; First posted 2012-07-10 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Healthy Participants
Keywords: Healthy participants; Hepatitis C virus; Telaprevir; Phenytoin; Carbamazepine; HCV; Interaction
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir; Phenytoin; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Panel 1 (Experimental): Part 1 of Panel 1: Participants will receive telaprevir 750 mg every 8 hours from Day 1 to Day 9 followed by a single 750-mg dose in the morning on Day 10. Part 2 of Panel 1: Participants will receive phenytoin 200 mg every 12 hours from Day 1 to Day 16 followed by a single 200-mg dose in the morning on Day 17; and telaprevir 750 mg every 8 hours from Day 8 to Day 16 followed by a single 750-mg dose in the morning on Day 17.
  Interventions: Drug: Telaprevir; Drug: Phenytoin
- Panel 2 (Experimental): Part 1 of Panel 2: Participants will receive telaprevir 750 mg every 8 hours from Day 1 to Day 9 followed by a single 750-mg dose in the morning on Day 10. Part 2 of Panel 2: Participants will receive carbamazepine 200 mg every 12 hours from Day 1 to Day 16 followed by a single 200-mg dose in the morning on Day 17; and telaprevir 750 mg every 8 hours from Day 8 to Day 16 followed by a single 750-mg dose in the morning on Day 17.
  brief description of the arm. This element may not be necessary if the associated intervention descriptions contain sufficient information to describe the arm.
  Interventions: Drug: Telaprevir; Drug: Carbamazepine

INTERVENTIONS:
Drug: Telaprevir — Type=exact number, unit=mg, number=375, form=tablet, route=oral. Two tablets of telaprevir will be administered as per the dosing regimens for each part of both the panels.
Drug: Phenytoin — Type=exact number, unit=mg, number=100, form=capsule, route=oral. Two capsules of phenytoin will be administered as per the dosing regimen in Part 2 of Panel 1.
  Arms: Panel 1
Drug: Carbamazepine — Type=exact number, unit=mg, number=200, form=tablet, route=oral. One tablet of carbamazepine will be administered as per dosing regimen in Part 2 of Panel 2.
  Arms: Panel 2

SUMMARY:
The purpose of this study is to investigate the potential pharmacokinetic (what the body does to the drug) interactions between multiple doses of phenytoin 200 mg every 12 hours or carbamazepine 200 mg every 12 hours and telaprevir 750 mg every 8 hours at steady-state (constant concentration of medication in the blood) in healthy participants.

DETAILED DESCRIPTION:
This is a Phase I, open-label (all people know the identity of the intervention), randomized (the study medication is assigned by chance), 2-panel, sequential treatment study. In this study 24 healthy participants will be randomly assigned equally to 2 panels. In Panel 1 the participants will receive telaprevir in Part 1 (telaprevir 750 mg every 8 hours from Day 1 to Day 9 followed by a single 750 mg dose in the morning on Day 10) and phenytoin/telaprevir in Part 2 (phenytoin 200 mg every 12 hours from Day 1 to Day 16 followed by a single 200-mg dose in the morning on Day 17; and telaprevir 750 mg every 8 hours from Day 8 to Day 16 followed by a single 750 mg dose in the morning on Day 17). In Panel 2 the participants will receive telaprevir (telaprevir 750 mg every 8 hours from Day 1 to Day 9 followed by a single 750 mg dose in the morning on Day 10) and carbamazepine/ telaprevir (carbamazepine 200 mg every 12 hours from Day 1 to Day 16 followed by a single 200-mg dose in the morning on Day 17; and telaprevir 750 mg every 8 hours from Day 8 to Day 16 followed by a single 200-mg dose in the morning on Day 17). In both panels, Part 1 and Part 2 are separated by a washout period of at least 2 weeks and maximum 4 weeks. Safety and tolerability will be assessed by evaluating adverse events, electrocardiogram, clinical laboratory examinations, vital signs and physical examination throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy on the basis of physical examination, medical history, vital signs, clinical laboratory tests, and electrocardiogram performed at screening
* If a woman, before entry she must be postmenopausal for at least 2 years (amenorrheal for at least 3 years), or surgically sterile (have had a total hysterectomy or bilateral oophorectomy, tubal ligation/bilateral tubal clips without reversal operation, or otherwise be incapable of becoming pregnant)
* Men must agree to use a highly effective method of birth control (ie, male condom with either female intrauterine device [IUD], diaphragm, cervical cap or hormone based contraceptives by their female partner) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* A 12-lead electrocardiogram consistent with normal cardiac conduction and function

Exclusion Criteria:

* Participants with a history of any illness that, in the opinion of the Investigator or the participant's general practitioner, might confound the results of the study or pose an additional risk in administering study drug(s) to the participant
* Participants of Asian ancestry (given association of phenytoin / carbamazepine and severe rash with HLA-B 1502 in this population)
* Current use of prescription medication, and regular use or routine use of concomitant medication(s), including over-the-counter (OTC) products
* Consumption of herbal medications or dietary supplements (eg, St. John's Wort, Ginkgo biloba, garlic supplements), vitamins, and grapefruit or grapefruit juice, apple juice, or orange juice within 14 days before the first administration of study drug
* Consumption of an average of more than five 240-mL servings of coffee or other caffeinated beverage per day

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Observed maximum plasma concentration (Cmax) of telaprevir. | Part 1: predose (Day 1, 8, 9 , and 10) and post dose 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, and 8h(Day 1 and Day 10); Part 2: predose (Day 1, 2, 6, 7, 8, 9, 10, 15, 16, and 17) and post dose 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, 8h, and 12h (Day 7, 8, and 17)
Area under the plasma concentration time curve from time of administration up to 8 hours post dose (AUC8h) of telaprevir. | Part 1: predose (Day 1, 8, 9 , and 10) and post dose 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, and 8h(Day 1 and Day 10); Part 2: predose (Day 1, 2, 6, 7, 8, 9, 10, 15, 16, and 17) and post dose 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, 8h, and 12h (Day 7, 8, and 17)
Observed minimum plasma concentration (Cmin) of telaprevir. | Part 1: predose (Day 1, 8, 9 , and 10) and post dose 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, and 8h(Day 1 and Day 10); Part 2: predose (Day 1, 2, 6, 7, 8, 9, 10, 15, 16, and 17) and post dose 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, 8h, and 12h (Day 7, 8, and 17)
Observed maximum plasma concentration (Cmax) of carbamazepine. | Part 1: predose (Day 1, 8, 9 , and 10) and post dose 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, and 8h(Day 1 and Day 10); Part 2: predose (Day 1, 2, 6, 7, 8, 9, 10, 15, 16, and 17) and post dose 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, 8h, and 12h (Day 7, 8, and 17)
Area under the plasma concentration time curve from time of administration up to 12 hours post dose (AUC12) of carbamazepine. | Part 1: predose (Day 1, 8, 9 , and 10) and post dose 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, and 8h(Day 1 and Day 10); Part 2: predose (Day 1, 2, 6, 7, 8, 9, 10, 15, 16, and 17) and post dose 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, 8h, and 12h (Day 7, 8, and 17)
Observed minimum plasma concentration (Cmin) of carbamazepine. | Part 1: predose (Day 1, 8, 9 , and 10) and post dose 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, and 8h(Day 1 and Day 10); Part 2: predose (Day 1, 2, 6, 7, 8, 9, 10, 15, 16, and 17) and post dose 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, 8h, and 12h (Day 7, 8, and 17)
Observed maximum plasma concentration (Cmax) of phenytoin. | Part 1: predose (Day 1, 8, 9 , and 10) and post dose 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, and 8h(Day 1 and Day 10); Part 2: predose (Day 1, 2, 6, 7, 8, 9, 10, 15, 16, and 17) and post dose 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, 8h, and 12h (Day 7, 8, and 17)
Area under the plasma concentration time curve from time of administration up to 12 hours post dose (AUC12) of phenytoin. | Part 1: predose (Day 1, 8, 9 , and 10) and post dose 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, and 8h(Day 1 and Day 10); Part 2: predose (Day 1, 2, 6, 7, 8, 9, 10, 15, 16, and 17) and post dose 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, 8h, and 12h (Day 7, 8, and 17)
Observed minimum plasma concentration (Cmin) of phenytoin. | Part 1: predose (Day 1, 8, 9 , and 10) and post dose 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, and 8h(Day 1 and Day 10); Part 2: predose (Day 1, 2, 6, 7, 8, 9, 10, 15, 16, and 17) and post dose 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, 8h, and 12h (Day 7, 8, and 17)

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to Day 17
Number of participants with abnormal values of laboratory results | Up to Day 17
Number of participants with abnormal electrocardiogram values | Up to Day 17
Number of participants with abnormal pulse and blood pressure values | Up to Day 17
Number of patients with abnormal physical examination findings | Up to Day 17

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Infectious Diseases BVBA Clinical Trial, Study Director — Janssen Infectious Diseases BVBA
Locations (1):
- Groningen, Netherlands